CLINICAL TRIAL: NCT05454215
Title: Mechanical INsufflator/EXsufflator Technique in Paediatric Subjects With Neuromuscular Disease: a Randomised Crossover Comparison of 2 Modes of Application
Brief Title: Mechanical Insufflator/Exsufflator Technique in Children With Neuromuscular Disease
Acronym: MINEX-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MINEX-2
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Neuromuscular Diseases in Children
Keywords: Lung function

STUDY DESIGN:
Intervention Model Description: Single center non-blinded randomized crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional settings first, modified settings second (Active Comparator): The control intervention (CON) is the conventional mode of a commercially available mechanical insufflator/exsufflator. The manoeuvre consists of 5 sets of 5 mechanical insufflations/exsufflations with individual pressure settings.
  For the study, the same pressure settings will be used as during daily routine.
  The study intervention (MOD) is a modified mode of a commercially available mechanical insufflator/exsufflator in which the active exsufflation of the last breath of each set will be omitted. The manoeuvre consists of 5 sets of 5 mechanical insufflations/exsufflations with individual pressure settings.
  For the study, the same pressure settings will be used as during daily routine. This modified mode is already used in daily routine by a minority of subjects with NMD.
  Interventions: Device: Mechanical insufflation/exsufflation conventional; Device: Mechanical insufflation/exsufflation modified
- Modified settings first, conventional settings second (Experimental): The study intervention (MOD) is a modified mode of a commercially available mechanical insufflator/exsufflator in which the active exsufflation of the last breath of each set will be omitted. The manoeuvre consists of 5 sets of 5 mechanical insufflations/exsufflations with individual pressure settings.
  For the study, the same pressure settings will be used as during daily routine. This modified mode is already used in daily routine by a minority of subjects with NMD.
  The control intervention (CON) is the conventional mode of a commercially available mechanical insufflator/exsufflator. The manoeuvre consists of 5 sets of 5 mechanical insufflations/exsufflations with individual pressure settings.
  For the study, the same pressure settings will be used as during daily routine.
  Interventions: Device: Mechanical insufflation/exsufflation conventional; Device: Mechanical insufflation/exsufflation modified

INTERVENTIONS:
Device: Mechanical insufflation/exsufflation conventional — Conventional settings in a commercially available chest physiotherapy device
Device: Mechanical insufflation/exsufflation modified — Modified settings in a commercially available chest physiotherapy device

SUMMARY:
In a randomized cross-over design, two different modes of a mechanical insufflator/exsufflator applied to pediatric subjects with neuromuscular disease will be compared with respect to their short term effect on lung function, i.e. lung volume.

DETAILED DESCRIPTION:
At two consecutive regular outpatient clinic visits, each participant will perform a session of the insufflation/exsufflation technique.

Participants will be randomised by a computer-generated code to one of the two sequences (CON-MOD or MOD-CON) using sealed envelopes. The randomisation list will be generated by a study nurse of the Department of Paediatrics who is not a member of the study group.

The randomisation envelope will be opened by the treating physiotherapist immediately before the first treatment session.

Standardised intervention

At randomisation, the measurement belt of the EIT system will be fitted around the chest of the participant. Once correct fit is confirmed, the baseline measurement (T0) will be taken. After the baseline assessment, the participants will perform the conventional (CON) or modified (MOD) insufflator/exsufflator therapy session under supervision of a physiotherapist. In teh investigator's institution a therapy session consists of 5 series of 5 insufflation/exsufflation manoeuvres each (Cough assist E70, Philips Respironics, Hamburg, Germany). Positive and negative pressures will be set at the individual level of each subject.

Measurements Changes in lung volume and ventilation distribution will be assessed by electrical impedance tomography (EIT). These parameters will be obtained five minutes before (T0) and five, ten, twenty, forty and sixty minutes after the treatment session (T1 - T5). Measurements of 3 minutes will be recorded at each time point. Additionally EIT measurements will be performed continuously during the treatment session.

Electrical Impedance Tomography (EIT) is a non-invasive, radiation-free technique for the assessment of spatial and temporal ventilation distribution based on the changes in electrical properties of the tissue during the respiratory cycle. EIT measurements will be performed using a commercially available setup (PulmoVista 500, Draeger, Germany). Image reconstruction will be performed with the GREIT-algorithm using the torso mesh function. [Adler, 2009] Relative change in end-expiratory lung impedance (EELI) and the global inhomogeneity (GI) index, a measure of ventilation inhomogeneity, will be calculated using customized software (Matlab® R2021b, The MathWorks Inc., Nattick, MA, USA).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of a NMD
* Functional status: non-ambulatory
* Age >5 years and < 16 years
* Able to cooperate
* Daily home-use of cough assist as reported by the caregivers
* Written informed consent by the subject/caregiver

Exclusion Criteria:

* Acute respiratory infection at two consecutive outpatient clinic visits (marked increase in cough, change in sputum amount or colour, fever or malaise)
* Oxygen dependency (defined as need for oxygen to achieve a transcutaneous oxygen saturation of ≥92%)
* Skin lesions at the chest (preventing EIT measurements)
* Chest deformation preventing EIT measurements

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-07 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Change in end-expiratory lung impedance from baseline | 3-5 Minutes
  Change of end-expiratory lung volume estimated by electrical impedance tomography from baseline to immediately after a session of mechanical insufflation/exsufflation.

SECONDARY OUTCOMES:
Change in ventilation distribution from baseline | 3-5 Minutes
  Differences in ventilation distribution assessed with electrical impedance tomography from baseline to immediately after a session of mechanical insufflation/exsufflation.
Duration of effect | 15-20 minutes
  Duration of the postulated effect on lung volume assessed by electrical impedance tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Riedel, MD, Study Director — Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing upon request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Available from time of publication for up to two years
Access Criteria: email: thomas.riedel@insel.ch

REFERENCES:
- [Background] Casaulta C, Messerli F, Rodriguez R, Klein A, Riedel T. Changes in ventilation distribution in children with neuromuscular disease using the insufflator/exsufflator technique: an observational study. Sci Rep. 2022 Apr 29;12(1):7009. doi: 10.1038/s41598-022-11190-z. PMID 35488044